CLINICAL TRIAL: NCT06565039
Title: The SUPPORT CE Study: A Safety and Effectiveness Study of the SUpira System in Patients Undergoing High-Risk Percutaneous COronaRy InTervention (HRPCI)
Brief Title: A Safety and Effectiveness Study of the Supira System in Patients Undergoing HRPCI - CE Study
Acronym: SUPPORT CE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never submitted to any Ethics Committee, Competant Authorities or any regulatory body. It was decided to cancel the study and not to proceed.
Sponsor: Supira Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-10006
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ventricular Assist Device

STUDY DESIGN:
Intervention Model Description: The study is a prospective, non-randomized, single-arm, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Supira System (Experimental): Ventricular support indicated for use during elective or urgent high-risk percutaneous coronary interventions.
  Interventions: Device: Supira System

INTERVENTIONS:
Device: Supira System — The Supira System is a minimally invasive, miniaturized percutaneous ventricular assist (pVAD) system that is intended to provide temporary (≤4 hours) hemodynamic support to patients undergoing a high-risk percutaneous coronary intervention (HRPCI). The Catheter is inserted percutaneously via the femoral artery, across the aortic valve, and into the left ventricle under fluoroscopic guidance, with a portion remaining in the ascending aorta. The left ventricle is unloaded by pumping blood from the ventricle into the ascending aorta and systemic circulation.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of utilizing the Supira System to provide hemodynamic support during HRPCI.

DETAILED DESCRIPTION:
The Supira System is a temporary (≤ 4 hours) ventricular support device indicated for use during elective or urgent high-risk percutaneous coronary interventions (HRPCI) performed in hemodynamically stable patients with severe coronary artery disease when a heart team, including a cardiac surgeon, has determined HRPCI is the appropriate therapeutic option.

Use of the Supira System in these patients may prevent hemodynamic instability which can result from repeat episodes of reversible myocardial ischemia that occur during planned temporary coronary occlusions and may reduce peri- and postprocedural adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤90 years
2. Hemodynamically stable and will undergo elective or urgent (not emergent) HRPCI, where hemodynamic support is deemed necessary as determined by the institutional Heart Team.
3. Informed consent granted by the patient or legally authorized representative

Exclusion Criteria:

1. Cardiogenic shock or acutely decompensated pre-existing chronic heart failure a. Note: Cardiogenic shock is defined as: systemic hypotension (systolic blood pressure [BP] <90 mmHg or the need for inotropes/pressors to maintain a systolic BP >90 mmHg) plus one of the following: any requirement for inotropes/pressors prior to arrival at the catheterization laboratory, clinical evidence of end-organ hypoperfusion or use of IABP or any other circulatory support device at time of screening.
2. Stroke within 6 months of the index procedure, or any prior stroke with permanent neurologic deficit
3. Evidence of left ventricular thrombus as assessed by Transthoracic Echocardiogram (TTE)
4. Aortic valvular disease or regurgitation categorized as moderate or greater (≥ 2+ on a 4-grade scale as assessed on TTE)
5. Aortic valve stenosis categorized as moderate or greater (gradient >20 mmHg or valve area <1.5 cm2 as assessed on TTE)
6. Previous aortic valve replacement or repair
7. Ascending or descending aortic dissection or aortic aneurysm >4.5 cm
8. Aortic and iliofemoral anatomical conditions that preclude safe delivery and placement of the investigational device
9. Presence of decompensated liver disease; severe liver dysfunction (Child class C)
10. Ongoing renal replacement therapy with dialysis
11. Infection of the proposed procedural access site or active systemic infection requiring ongoing antibiotic therapy
12. Heparin-induced thrombocytopenia, current or any prior occurrences
13. Known hypersensitivity to intravenous contrast agents that cannot be adequately pre-medicated or known hypersensitivity to heparin, aspirin, adenosine diphosphate (ADP) receptor inhibitors, or nitinol
14. Known or suspected coagulopathy or abnormal coagulation parameters (defined as platelet count ≤ 100,000/mm³ or spontaneous International Normalized Ratio (INR) ≥ 1.5 or known fibrinogen ≤ 1.5 g/L)
15. Any condition or scheduled surgery that will require discontinuation of antiplatelet and/or anticoagulant therapy within 90 days of the index procedure
16. Planned coronary intervention within 30 days prior or post index procedure
17. Breastfeeding or pregnant or planning to become pregnant within 90 days of the HRPCI procedure
18. Currently participating in active follow-up phase of another clinical study of an investigational drug or device or planning to enroll in such a study within 90 days of the HRPCI procedure
19. Active COVID-related infection or prior COVID-19 diagnosis with sequelae that could confound endpoint assessments
20. Other medical, social, or psychological problems that would have them be considered in any way to be part of a vulnerable population. This includes individuals who may have difficulty providing informed consent or are at a higher risk of coercion or undue influence, individuals permanently incapable of giving informed consent, and individuals whose ability to comply with study procedures may be compromised, in the opinion of the Investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Successful initiation and maintenance of hemodynamic support | 90 days from procedure
  A composite endpoint of safety and effectiveness outcomes, evaluated at 90 days, comprises the following outcomes:
  * All-cause death
  * Myocardial infarction (MI)
  * Stroke or transient ischemic attack (TIA)
  * Unplanned repeat revascularization
  * Major bleeding (BARC ³ 3)
  * Major vascular complications (MCS-ARC defined)
  * Sustained hypotension during mechanical circulatory support

SECONDARY OUTCOMES:
Procedural Success | 90 days from procedure
  Freedom from:
  1. Major bleeding (BARC ³ 3)
  2. Major vascular complications (MCS-ARC defined)
  3. Sustained hypotension during mechanical circulatory support
  4. Need for mechanical circulatory support beyond the index procedure

IPD SHARING:
Plan to Share IPD: No